CLINICAL TRIAL: NCT05663645
Title: Navigating Health Insurance Selection for in Vitro Fertilization (IVF) Benefits
Brief Title: Navigating Health Insurance Selection for IVF Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Hui-Chun Irene Su, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 805955
Record Dates: First submitted 2022-12-01; First posted 2022-12-23 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Infertility
Keywords: infertility; IVF; health insurance
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health insurance educational guide (Experimental): Eligible individuals will receive a health insurance educational guide to support choosing among 5 health plans for IVF coverage. They will also receive receive a one-page guide with a link to the Open Enrollment website that is available to all employees during the open enrollment period.
  Interventions: Behavioral: Health insurance educational guide
- Usual care (No Intervention): Eligible individuals will receive a one-page guide with a link to the Open Enrollment website that is available to all employees during the open enrollment period.

INTERVENTIONS:
Behavioral: Health insurance educational guide — The educational guide includes 4 content areas: 1) Definition of key insurance terms; 2) premiums, deductibles across the five 2023 health plans; 3) Summary of how premiums and deductibles can affect out of pocket costs; 4) Guide to finding in-network IVF providers and facilities.
  Arms: Health insurance educational guide

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an educational intervention on health insurance literacy and utilization of in vitro fertilization (IVF) insurance benefits. The investigators hypothesize that the intervention is acceptable and satisfactory and will result in increased health insurance literacy and utilization of IVF benefits.

ELIGIBILITY:
Inclusion Criteria:

* Employees eligible for health insurance coverage
* Reproductive aged (18 to 50 years)
* Intention to grow their family in the next year
* Primary language English or Spanish

Exclusion Criteria:

* None

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Health Insurance Literacy Measure | 10 months after receipt of the intervention
  9 items from the Health Insurance Literacy Measure will assess participants' confidence using their health insurance and being proactive with their health insurance for IVF services. Items will be scored from 0 (not at all confident) to 3 (very confident). Higher scores indicate better health insurance literacy.

SECONDARY OUTCOMES:
Health Insurance Literacy Measure | 1 month after receipt of the intervention
  6 items from the Health Insurance Literacy Measure will assess participants' likelihood of comparing health insurance plans. Items will be scored from 0 (not at all confident) to 3 (very confident). Higher scores indicate better health insurance literacy.
Utilization of IVF services | 10 months after receipt of the intervention
  Participants will self-report utilization of IVF services.
Insurance coverage | 10 months after receipt of the intervention
  Participants will self-report insurance coverage related to IVF services.
Out of pocket expenses | 10 months after receipt of the intervention
  Participants will self-report out-of-pocket expenses related to IVF services.
Financial hardship | 10 months after receipt of the intervention
  The 15-item Economic Strain and Resilience in Cancer tool will be used as a self-report subjective measure of financial hardship related to infertility and IVF services. Items are scored from 0 (least hardship) to 10 (most severe hardship). Higher scores indicate worse financial hardship.

CONTACTS AND LOCATIONS:
Overall Officials: H. Irene Su, MD MSCE, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data generated during the study will be available from the principal investigator (H. Irene Su) upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication.
Access Criteria: Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to the principal investigator (H. Irene Su).

REFERENCES:
- [Derived] Dayo O, Turcotte V, Reyes B, Flores Ortega RE, Kaiser BN, Aarons GA, McMenamin SB, Su HI, Romero SAD. Navigating health insurance selection for in vitro fertilization (IVF) benefits: A study protocol. Contemp Clin Trials. 2025 Aug;155:107998. doi: 10.1016/j.cct.2025.107998. Epub 2025 Jun 30. PMID 40602660